CLINICAL TRIAL: NCT06422845
Title: A Prospective, Multicenter, Single-Arm Target Value Clinical Study to Evaluate the Safety and Effectiveness of Peripheral Scoring Drug-coated Balloon Dilation Catheter in the Treatment of Hemodialysis Arteriovenous Fistula Stenosis
Brief Title: Peripheral Scoring Drug-coated Balloon in the Treatment of Hemodialysis Arteriovenous Fistula Stenosis
Acronym: SCDB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DK Medical Technology (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-P-24-012
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Arteriovenous Fistula Stenosis
Keywords: arteriovenous fistula stenosis; scoring; hemodialysis; drug-coated balloon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dissolve AV Peripheral Scoring Drug-coated Balloon (Experimental): Subjects in this group are treated with Dissolve AV Peripheral Scoring Drug-coated Balloon dilatation catheter
  Interventions: Device: Dissolve AV Peripheral Scoring Drug-coated Balloon

INTERVENTIONS:
Device: Dissolve AV Peripheral Scoring Drug-coated Balloon — Subjects in the test group are treated with Dissolve AV Peripheral Scoring Drug-coated Balloon
  Other Names: Scoring Drug-coated Balloon

SUMMARY:
This is a prospective, multi-center, single-arm target value clinical study to study the safety and effectiveness of Peripheral Scoring Drug-coated Balloon dilatation catheters in the treatment of hemodialysis arteriovenous fistula stenosis.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm target value clinical study to study the safety and effectiveness of Peripheral Scoring Drug-coated Balloon dilatation catheters (SDCB) in the treatment of hemodialysis arteriovenous fistula stenosis. A total of 328 participants will be enrolled across multiple clinical trial sites. Participants will undergo a surgical procedure using a peripheral scoring drug-coated balloon dilation catheter, with follow-up within 5 days, at 1 month, and 6 months after the procedure, then at 12, 18, and 24 months post-procedure. The target lesion primary patency (TLPP) at 6 months post-procedure is the defined primary endpoint to evaluate the safety and effectiveness of the peripheral scoring drug balloon dilatation catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years old;
2. The patient's AVF/AVG is mature and has successfully completed hemodialysis at least once;
3. The target lesion is located at the AVF/AVG return vein and venous side anastomosis;
4. Hemodynamically significant AVF/AVG return vein stenosis ≥ 50% as assessed by ultrasound or contrast imaging, and any of the following clinical symptoms, signs or indicators are present, including significant increase in venous pressure during dialysis, abnormal physical examination, decreased pump-controlled blood flow, decreased adequacy of dialysis, brachial artery blood flow < 600 ml/min or decreased by 25% compared with the previous follow-up visit, etc.;
5. The target lesion is a primary or restenotic lesion, consisting of one or more tandem lesions (if the total length of adjacent tandem lesions is ≤ 60 mm, it can be considered a single target lesion);
6. Visual inspection of the reference blood vessel diameter of the target lesion is between 4.0-8.0mm, and the total length of the target lesion is ≤ 60mm;
7. The patient voluntarily signs the informed consent form.

Exclusion Criteria:

1. Women of childbearing age whose preoperative pregnancy test is not negative, and women who are breastfeeding;
2. Patients who have undergone major surgical treatment within 30 days before inclusion in the study;
3. Calcified lesions that are not expected to be expandable with balloons;
4. Patients with thrombosis at the access stenosis site;
5. The target lesion is located at the blood supply artery and arterial anastomosis;
6. Patients known to be allergic to or intolerant to contrast media and paclitaxel;
7. The patient's life expectancy is less than 2 years;
8. Patients with systemic lupus erythematosus and antineutrophil cytoplasmic antibody (ANCA)-associated small vessel vasculitis;
9. Patients with kidney transplantation or those who planned to undergo kidney transplantation or switch to peritoneal dialysis;
10. Vascular access infection or systemic active infection;
11. Those who have participated in unfinished clinical trials of other drugs or devices;
12. Patients with other medical conditions that the investigator believes are not suitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Primary Patency (TLPP) at 6 months post-procedure | 6 months post-procedure
  Target Lesion Primary Patency is defined as freedom from clinically driven Target Lesion Failure (TLF) (including +/-5mm proximal or distal of the target lesion) or Vascular Access Thrombosis.
  TLF is defined as the presence of at least one clinical symptom, sign or indicator (defined according to the NKF-K/DOQI guideline) due to target lesion stenosis (≥ 50% stenosis of the target lesion assessed by contrast angiography or ultrasound), including a significant increase in venous pressure during dialysis, high blood pressure, abnormal physical examination, decreased pump-controlled blood flow, decreased dialysis adequacy, brachial artery blood flow < 600 ml/min or decreased by 25% compared with the previous follow-up, etc.

SECONDARY OUTCOMES:
Target Lesion Primary Patency (TLPP) | 12, 24 months post-procedure
  TLF is defined as the presence of at least one clinical symptom, sign or indicator (defined according to the NKF-K/DOQI guideline) due to target lesion stenosis (≥ 50% stenosis of the target lesion assessed by contrast angiography or ultrasound), including a significant increase in venous pressure during dialysis, high blood pressure, abnormal physical examination, decreased pump-controlled blood flow, decreased dialysis adequacy, brachial artery blood flow < 600 ml/min or decreased by 25% compared with the previous follow-up, etc.
Proportion of patients whose peak systolic flow velocity ratio (PSVR) ≤ 2.0, as determined by Doppler ultrasound (DUS), so as to confirm the absence of restenosis | 6, 12, 24 months post-procedure
  Proportion of patients whose peak systolic flow velocity ratio (PSVR) ≤ 2.0, as determined by Doppler ultrasound (DUS), at 6, 12, and 24 months post-procedure, so as to confirm the absence of restenosis.
Clinically-driven Target Lesion Revascularization (CD-TLR) | 1, 6, 12, 18, and 24 months post-procedure
  Any reintervention of a target lesion (including +/-5 mm proximal or distal to the target lesion) as determined by clinical symptoms or dialysis indicators indicating that it is unable to perform dialysis.
Clinically-driven Target Shunt Revascularization (CD-TSR) | 1, 6, 12, 18, and 24 months post-procedure
Device Success | During the procedure
  Defined as the ability of the balloon to reach the target lesion, be successfully expanded without rupture, and be successfully withdrawn. Evaluation is based on single balloon dilation catheter.
Technical Success | 0-5 days post-procedure
  Defined as residual stenosis of the target lesion post-procedure is ≤ 30%, and no serious adverse events related to the trial device occurred during the perioperative period.
Clinical Success | 0-5 days post-procedure
  Defined as ability to complete at least one successful hemodialysis session post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Yuzhu Wang, MD, Principal Investigator — Beijing Haidian Hospital
Locations (33):
- China (33):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Haidian Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou First People's Hospital, Guanzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Eighth Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong
  - Liuzhou Traditional Chinese Medical Hospital, Liuchow, Guangxi
  - Foresea Life Insurance Guangxi Hospital, Nanning, Guangxi
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated To Tongji Medical College HUST, Wuhan, Hubei
  - Changsha Jieao Kidney Disease Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Affiliated Hospital To Changchun University of Chinese Medicine, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University Dezhou Hospital, Dezhou, Shandong
  - Central Hospital Affiliated To Shandong First Medical University, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - People's Hospital of Rizhao, Rizhao, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Sir Run Run Shaw Hospital Zhejiang University School of medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jinhua Hospital of TCM, Jinhua, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Ürümqi

IPD SHARING:
Plan to Share IPD: No